CLINICAL TRIAL: NCT03286049
Title: Short and Mid-term Repeatability of Active Anterior Rhinomanometry (AAR) Measurements in Paediatric Age - Rhino-Rep
Brief Title: Short and Mid-term Repeatability of Active Anterior Rhinomanometry (AAR) Measurements in Paediatric Age
Acronym: Rhino-Rep
Status: Completed | Type: Observational
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Ph.D. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: 7/2017_C
Record Dates: First submitted 2017-09-05; First posted 2017-09-18 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Rhinitis; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic; Rhinitis, Allergic, Seasonal; Rhinitis, Allergic, Perennial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy children (HC): 10 healthy children
- Children with non allergic rhinitis (NAR): 10 children with non allergic rhinitis
- Rhinitis children, perennial allergy (PAR): 10 rhinitis children, sensitized to perennial allergens
- Rhinitis children, seasonal allergy, outside season (OSR): 10 rhinitis children sensitized to seasonal allergens, observed outside the allergen season
- Rhinitis children, seasonal allergy, within season (WSR): 10 rhinitis children sensitized to seasonal allergens, observed during the allergen season

SUMMARY:
Longitudinal, observational study to assess the short-term (test re-test) and mid-term (within the span of 28 days) repeatability of active anterior rhinomanometry (AAR) measures on 4 parallel groups of children with different rhinitis phenotypes, and 1 group of control (healthy) children.

Secondary objectives are: i) assessing of association between AAR, exhaled FeNO (eFeNO) and nasal FeNO (nFeNO); ii) assessing association between objective measurements (AAR, eFeNO and nFeNO) and subjective measurements (Total 5 Symptom score, T5SS).

The study is intended to obtain useful information for improving rhinitis management.

ELIGIBILITY:
Healthy volunteers (HC)

The inclusion criteria for HC are:

1. Negative bronchodilator response;
2. No major nasal septum malformations.

The exclusion criteria for HC are:

1. Upper airway infections in the previous 4 weeks;
2. Active smoker;
3. Lifetime history of asthma, rhinitis, or respiratory disease symptoms.

Children with non allergic rhinitis (NAR)

The inclusion criteria for NAR are:

1.T5SS>5 in the last 4 weeks.

The exclusion criteria for NAR are:

1. At least one positive skin prick test for aeroallergens;
2. Upper airway infections in the previous 4 weeks;
3. Active smoker;
4. Major nasal septum malformations.

Rhinitis children, perennial allergy (PAR)

The inclusion criteria for PAR are:

1. T5SS>5 in the last 4 weeks.
2. At least one positive skin prick test for perennial aeroallergens;

The exclusion criteria for PAR are:

1. At least one positive skin prick test for seasonal aeroallergens;
2. Upper airway infections in the previous 4 weeks;
3. Active smoker;
4. Major nasal septum malformations.

Rhinitis children, seasonal allergy, outside season (OSR)

The inclusion criteria for OSR are:

1. T5SS>5 in the last 4 weeks.
2. At least one positive skin prick test for seasonal aeroallergens;

The exclusion criteria for OSR are:

1. At least one positive skin prick test for perennial aeroallergens;
2. Upper airway infections in the previous 4 weeks;
3. Active smoker;
4. Major nasal septum malformations.

Rhinitis children, seasonal allergy, within season (OSR)

The inclusion criteria for OSR are:

1. T5SS>5 in the last 4 weeks.
2. At least one positive skin prick test for seasonal aeroallergens;

The exclusion criteria for OSR are:

1. At least one positive skin prick test for perennial aeroallergens;
2. Upper airway infections in the previous 4 weeks;
3. Active smoker;
4. Major nasal septum malformations.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A study population of 40 rhinitis children (10 for each of 4 different rhinitis phenotypes)
  attending the outpatient clinic of Pediatric Allergology & Pulmonology (PAP) within the Institute
  of Biomedicine and Molecular Immunology (IBIM) of the National Research Council (CNR) of Palermo (IBIM CNR), and a control group of 10 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Short term repeatability of active anterior rhinomanometry (AAR) | 1 day
  For each individual, it will be calculated the coefficient of variation of 5 measurements of AAR taken within 30 minutes, at baseline.
Mid term repeatability of active anterior rhinomanometry (AAR) | 28 days
  For each individual, it will be calculated the coefficient of variation of 3 measurements of AAR taken at baseline and then twice more within the span of 28 days (after one week and after two weeks).

SECONDARY OUTCOMES:
Correlation between AAR and oral FeNO | 28 days
  Correlation coefficients between measurements of AAR and oral FeNO (at each visit the mean of 3 consecutive measurements of oral FeNO is considered)
Correlation between AAR and nasal FeNO | 28 days
  Correlation coefficients between measurements of AAR and nasal FeNO (at each visit the mean of 3 consecutive measurements of nasal FeNO is considered)
Correlation between AAR (objective perspective) and T5SS (subjective perspective) | 28 days
  Correlation coefficients between measurements of AAR and total 5 symptom score
Correlation between FeNO (objective perspective) and T5SS (subjective perspective) | 28 days
  Correlation coefficients between measurements of FeNO and total 5 symptom score

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM), National Research Council, Palermo, Sicily, Italy

REFERENCES:
- [Derived] Cilluffo G, Zicari AM, Ferrante G, Malizia V, Fasola S, Duse M, De Castro G, De Vittori V, Schiavi L, Brindisi G, Petrelli P, La Grutta S. Assessing repeatability and reproducibility of Anterior Active Rhinomanometry (AAR) in children. BMC Med Res Methodol. 2020 Apr 17;20(1):86. doi: 10.1186/s12874-020-00969-1. PMID 32303189